CLINICAL TRIAL: NCT04415827
Title: Study of Energy Supply in Athletes and Untrained Persons With Diseases of the Bronchopulmonary System
Brief Title: Energy Supply in Athletes and Untrained Persons With Bronchopulmonary Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 520122019
Record Dates: First submitted 2020-04-17; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Community-acquired Pneumonia; Bronchitis; Chronic Obstructive Pulmonary Disease; Acute Respiratory Infection
Keywords: sports medicine; bicycle ergometry; bronchopulmonary diseases; spiroergometry
MeSH Terms: conditions — Community-Acquired Pneumonia; Bronchitis; Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Athletes with community-acquired pneumonia (Experimental): man and women, athletes, age 17-25, patients with community-acquired pneumonia
  Interventions: Diagnostic Test: bicycle ergometry test with spiroergometry
- Untrained people with community-acquired pneumonia (Experimental): man and women, untrained people, age 17-25, patients with community-acquired pneumonia
  Interventions: Diagnostic Test: bicycle ergometry test with spiroergometry
- Athletes with bronchitis (Experimental): man and women, athletes, age 17-25, patients with bronchitis
  Interventions: Diagnostic Test: bicycle ergometry test with spiroergometry
- Untrained people with bronchitis (Experimental): man and women, untrained people, age 17-25, patients with bronchitis
  Interventions: Diagnostic Test: bicycle ergometry test with spiroergometry
- Athletes with chronic obstructive pulmonary disease (Experimental): man and women, athletes, age 17-25, patients with with chronic obstructive pulmonary disease
  Interventions: Diagnostic Test: bicycle ergometry test with spiroergometry
- Untrained people with chronic obstructive pulmonary disease (Experimental): man and women, untrained people, age 17-25, patients with with chronic obstructive pulmonary disease
  Interventions: Diagnostic Test: bicycle ergometry test with spiroergometry
- Athletes with acute respiratory infections (Experimental): man and women, athletes, age 17-25, patients with acute respiratory infections
  Interventions: Diagnostic Test: bicycle ergometry test with spiroergometry
- Untrained people with acute respiratory infections (Experimental): man and women, untrained people, age 17-25, patients with acute respiratory infections
  Interventions: Diagnostic Test: bicycle ergometry test with spiroergometry

INTERVENTIONS:
Diagnostic Test: bicycle ergometry test with spiroergometry — The 1st testing will be carried out on the 28-31th day of the disease, which corresponds to the period of the expected normalization of temperature, improvement of well-being, positive dynamics of radiological (with community-acquired pneumonia) and laboratory data, the 2nd test - after 3 months, the 3rd - after 6 months and IV - after 12 months.
  Load testing will be carried out on a bicycle ergometer with an initial power of 25 watts with a further increase of 25 watts every 3 minutes. The cessation of the load will be carried out upon the appearance of signs set forth in the recommendations of the World Health Organization Expert Committee (1970)

SUMMARY:
Study of the energy supply of bicycle ergometric load in athletes and untrained persons with bronchopulmonary diseases (community-acquired pneumonia, bronchitis, chronic obstructive pulmonary disease and acute respiratory viral infections, to justify the timing of the resumption of training, as well as determination of the volume and intensity of physical activity in training and competitive processes.

DETAILED DESCRIPTION:
1. The aim of the study is to assess energy supply of bicycle ergometric load in athletes and untrained persons who have suffered diseases of the bronchopulmonary system (community-acquired pneumonia, bronchitis, chronic obstructive pulmonary disease and acute respiratory viral infections, to justify the timing of the resumption of training, as well as determining the volume and the intensity of physical activity in the training and competitive processes.
2. In addition to a comprehensive general clinical, radiological (for community-acquired pneumonia) and laboratory examination, all the subjects under study will undergo special studies: spirography and spiroergometry, electrocardiography (ECG), and bicycle ergometry.
3. The main indicators of the functional state of the cardio-respiratory system of the study participants are indicators of the function of external respiration and gas exchange, recorded in the initial state, after load and in the recovery period of 10 and 30 minutes.

Patients with diseases of the bronchopulmonary system will receive treatment according to generally accepted standards of drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. the presence of written informed consent of the patient to participate in the study;
2. athletes (men and women) with a diagnosis of community-acquired pneumonia / bronchitis / chronic obstructive pulmonary disease / acute respiratory viral infection on days 28-31 from the onset of the disease, i.e. in the stage of clinical recovery;
3. untrained individuals (men and women) with a diagnosis of community-acquired pneumonia / bronchitis / chronic obstructive pulmonary disease / acute respiratory viral infection;
4. age 17 - 25 years.

Exclusion Criteria:

1. refusal of the patient from further participation in the study;
2. non-compliance with treatment recommendations and regimen.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-05-23 (Actual); Primary Completion 2021-12-22 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of the respiratory system function at different periods of the bronchopulmonary disease | The 1st test will be carried out on the 28-31th day of the disease, the 2nd test - after 3 months, III - after 6 months and IV - after 12 months.
  assesment a change of respiratory rate using stress test machine "Cardiovit" in the initial state, after cycling and in the recovery period for 10 and 30 minutes.
Change of the cardiovascular system function at different periods of the bronchopulmonary disease | The 1st test will be carried out on the 28-31th day of the disease, the 2nd test - after 3 months, III - after 6 months and IV - after 12 months.
  assesment a change of heart rate using stress test machine "Cardiovit" in the initial state, after cycling and in the recovery period for 10 and 30 minutes.

SECONDARY OUTCOMES:
Change of electrical activity of the heart at different periods of the bronchopulmonary disease | The 1st test will be carried out on the 28-31th day of the disease, the 2nd test - after 3 months, III - after 6 months and IV - after 12 months.
  assesment a change of the electrical activity of the heart using stress test machine "Cardiovit", recording changes on an ECG (segment ST) during cycling.
Change of pulmonary ventilation at different periods of the bronchopulmonary disease | The 1st test will be carried out on the 28-31th day of the disease, the 2nd test - after 3 months, III - after 6 months and IV - after 12 months.
  assesment a change of the pulmonary ventilation using stress test machine "Cardiovit", determining tidal volume (l/min) in the initial state, after cycling and in the recovery period for 10 and 30 minutes.
Change of pulmonary gas exchange at different periods of the bronchopulmonary disease | The 1st test will be carried out on the 28-31th day of the disease, the 2nd test - after 3 months, III - after 6 months and IV - after 12 months.
  assesment a change of oxygen uptake (ml/min) using stress test machine "Cardiovit" in the initial state, after cycling and in the recovery period for 10 and 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria S Moskvichyova, Study Chair — I.M. Sechenov First Moscow State Medical University
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
prohibited by Local Ethics Committee of "I.M. Sechenov First Moscow State Medical University"